CLINICAL TRIAL: NCT02148549
Title: The Pilot Study of Neoadjuvant Chemotherapy of FIRINOX for Patients With Borderline Resectable Pancreatic Cancer
Brief Title: Neoadjuvant FIRINOX for Borderline Resectable Pancreatic Cancer - a Pilot Study
Acronym: FIRINOX
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Wakayama Medical University (Other)
Responsible Party: Principal Investigator, Hiroki Yamaue, Dean & Professor, Wakayama Medical University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: FIRINOX; UMIN000013809 (Other: UMIN)
Record Dates: First submitted 2014-05-15; First posted 2014-05-28 (Estimated); Last update posted 2019-10-07 (Actual); Status verified 2015-07

CONDITIONS: Patients With Borderline Resectable Pancreatic Cancer
Keywords: Borderline resectable pancreatic cancer; R0 resection; Resection rate; Optimal schedule
MeSH Terms: interventions — Oxaliplatin; Irinotecan; Fluorouracil

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Optimal chemotherapy courses (Experimental): Neoadjuvant chemotherapy 4 courses of FIRINOX early 5 patients, and 8 courses of FIRINOX subsequent 5 patients
  Interventions: Drug: FIRINOX

INTERVENTIONS:
Drug: FIRINOX — FIRINOX regimen by eliminating LV and bolus 5-FU, and irinotecan reduced to 150mg/m2 of 180mg/m2 from FOLFIRINOX regimen.
  Other Names: Oxaliplatin, Irinotecan, 5-FU.

SUMMARY:
FOLFIRINOX regimen was recently presented at an international oncology meeting and represents a new standard regimen in the treatment of metastatic pancreatic cancer. FOLFIRINOX is one of the high response rate treatment regimen , the investigators considered as a promising treatment as neoadjuvant chemotherapy . On the other hand , incidences of grade 3 or 4 neutropenia , febrile neutropenia and diarrhea were significantly higher in the FOLFIRINOX group compared with gemcitabine group. Therefore, it was decided to consider the balance of safety and efficacy as a preoperative chemotherapy, the investigators use the FIRINOX regimen by eliminating LV and bolus 5-FU, and irinotecan reduced to 150mg/m2 of 180mg/m2 from FOLFIRINOX regimen

DETAILED DESCRIPTION:
FOLFIRINOX regimen was recently presented at an international oncology meeting and represents a new standard regimen in the treatment of metastatic pancreatic cancer. FOLFIRINOX is one of the high response rate treatment regimen , the investigators considered as a promising treatment as neoadjuvant chemotherapy . On the other hand , incidences of grade 3 or 4 neutropenia , febrile neutropenia and diarrhea were significantly higher in the FOLFIRINOX group compared with gemcitabine group. Therefore, it was decided to consider the balance of safety and efficacy as a preoperative chemotherapy, the investigators use the FIRINOX regimen by eliminating LV and bolus 5-FU, and irinotecan reduced to 150mg/m2 of 180mg/m2 from FOLFIRINOX regimen. The investigators also evaluate the optimal treatment schedule of FIRINOX therapy as neoadjuvant chemotherapy, optimal duration between surgery and chemotherapy, R0 resection rate, and resection rate for borderline resectable pancreatic cancer.

ELIGIBILITY:
Inclusion Criteria:

* Pathologically proven invasive pancreatic ductal carcinoma
* Cases that meet the definition of borderline resectable pancreatic cancer 1) or 2)

  1. Definition of a borderline resectable pancreatic cancer is filledin NCCN guideline version 1.2014 pancreatic adenocarcinoma
  2. Patients indicated distal pancreatectomy with en bloc celiac axis resection
* PS (ECOG) 0-1
* ≧20 years old and < 75 years old
* First line treatment
* The following criteria must be satisfied in laboratory tests within 14 days of registration White blood cell count ≦12,000/mm3 Neutrophil count ≧1,500/mm3 Platelet count ≧100,000mm3 Total bilirubin <2.0mg/dL Serum Creatinine ≦upper limits of normal(ULN) AST, ALT≦2.5×ULN Albumin≧3.0g/dL Hemoglobin≧9.0g/dL
* Written informed consent to participate in this study

Exclusion Criteria:

* Severe drug hypersensitivity
* Multiple primary cancers within 5 years
* Severe infection
* With grade2 or more severe peripheral neuropathy
* With intestinal paralysys, ileus
* Interstitial pneumonia or pulmonary
* With uncontrollable pleural effusion or ascites
* Receiving atazanavir sulfate
* With uncontrollable diabetes
* With uncontrollable heart failure, angina, hypertension, arrhythmia
* With severe psychological symptoms
* With watery diarrhea
* Pregnant or lactating women, or women with known or suspected pregnancy
* Inappropriate patients for entry on this study in the judgment of the investigator
* With UGT1A1*28 and/or UGT1A1*6 polymorphisms

Ages: 20 Years to 74 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2014-04; Primary Completion 2017-02 (Actual); Study Completion 2017-02 (Actual)

PRIMARY OUTCOMES:
Number of participants with toxicity of FIRINOX therapy as neoadjuvant chemotherapy for borderline resectable pancreatic cancer. | Up to 30 weeks.
  Toxicities will be assessed according to Common Terminology Criteria for Adverse Events (CTCAE) 4.0.

SECONDARY OUTCOMES:
The resection rate of FIRINOX therapy as neoadjuvant chemotherapy for borderline resectable pancreatic cancer. | Up to 24 weeks.
The R0 resection rate of FIRINOX therapy as neoadjuvant chemotherapy for borderline resectable pancreatic cancer. | Up to 30 weeks.
The optimal treatment schedule of FIRINOX therapy as neoadjuvant chemotherapy for borderline resectable pancreatic cancer. | Up to 2 years.

CONTACTS AND LOCATIONS:
Overall Officials: Hiroki Yamaue, M.D., PhD, Principal Investigator — Wakayama Medical University
Locations (9):
- Japan (9):
  - Nagoya University, Nagoya, Aichi-ken
  - Kobe University, Kobe, Hyōgo
  - Nara Prefectual Medical University, Kashihara, Nara
  - Kansai Medical University, Hirakata, Osaka
  - Osaka University, Suita, Osaka
  - Hiroshima University, Hiroshima
  - Osaka City University, Osaka
  - Osaka Medical Center for Cancer and CVD, Osaka
  - Wakayama Medical University, Wakayama